CLINICAL TRIAL: NCT00931398
Title: Treatment of College Students With ADHD Using OROS Methylphenidate
Brief Title: Treatment of College Students With Attention-Deficit/Hyperactivity Disorder (ADHD) Using OROS Methylphenidate
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not initiated due to lack of funding by the sponsor
Sponsor: University of Pittsburgh (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Oscar Bukstein, MD, MPH / Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ConcertaATT4100
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate HCl (Concerta) (Experimental)
  Interventions: Drug: methylphenidate HCl (Concerta)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate HCl (Concerta) — Concerta 18 mg, 36 mg, 54 mg, and 72 mg q.am.
  Other Names: Concerta
  Arms: Methylphenidate HCl (Concerta)
Drug: Placebo — Matched placebo for all Concerta doses.
  Arms: Placebo

SUMMARY:
The purpose of the proposed study is to determine the effectiveness of methylphenidate HCl (Concerta) in college students with ADHD. This study will consist of 110 college students between the ages of 18 and 25 who are enrolled full-time in a local or junior college. The study consists of an 8-week double-blind, placebo-controlled trial of placebo versus methylphenidate HCl (Concerta®) followed by a 10-week extension of open label methylphenidate HCl (Concerta®).

DETAILED DESCRIPTION:
There are very few trials on drug efficacy and safety treatment performed specifically for college students with Attention-Deficit/Hyperactivity Disorder (ADHD). Although data based on the adult population can often be extrapolated and generalized to a college population, there are unique treatment demands for college students with ADHD that are not represented in day-to-day functioning of adults with ADHD. For example, although adults may be able to choose employment that capitalizes on their skill sets and tolerate ADHD-related deficits, all college students must manage intensive learning experiences in an environment that places unparalleled demands on higher order cognitive processes that are deficient with ADHD. In addition, it may be important to address the comorbidities that may be common among ADHD college students. This could range from eating disorders, depression or anxiety to alcoholism and drug abuse. For example, heavy drinking peaks in the college student years regardless of ADHD but the long-term course and underlying predispositions may be different among individuals with a history of ADHD (Molina et al., 2007). Although there are a few case studies, there are limited studies on ADHD and their comorbidities in college students perhaps because it may be a challenge to recruit a respectable sample size. Furthermore, it may be important to recognize that some college students never develop diagnosable ADHD symptoms as children, and that the signs may manifest themselves in a very harmful way during college when demands for academic rigor and organization reach their height. Given the juxtaposing conditions of academic demand, autonomy from parents, and increased opportunities for drug abuse, it becomes imperative to directly address treatment in this population. Much more research is left to be performed on this unique population of ADHD patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-25 years, inclusive
* DSM-IV diagnosis of ADHD (any subtype)
* Clinical Global Impressions scale (CGI)-Severity score of ≥4 ("Moderately ill" or higher) for ADHD

Exclusion Criteria:

* Pregnancy or a history of seizure disorder, other neurological or medical disorder for which medication treatment may present a considerable risk
* Abnormal liver function
* History of pervasive developmental disorder, schizophrenia, other psychotic disorders, or eating disorders
* Currently taking other psychotropic medications from which discontinuation would present a significant risk (we will not allow subjects with a satisfactory medication response to discontinue that medication and to participate)
* Active substance dependence or lack of control of substance use that does not allow for safe medication administration

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy measures will be the self-reported CAARS DSM-IV ADHD Symptoms Total and the CAARS Inattention/Memory Problems indices (Connors et al., 1999) | 8 weeks

SECONDARY OUTCOMES:
Secondary measures include CAARS subscales, Barkley Adult ADHD Rating Scale, Impairment Rating Scale, General Life Functioning, final grades and GPA, substance use and associated negative consequences. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Bukstein, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Youth and Family Research Program, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: study site web page — http://www.youthandfamilyresearch.com